

Approved by the Human Subjects Ethics Sub-committee of The Hong Kong Polytechnic University on 13/04/2018





## CONSENT TO PARTICIPATE IN RESEARCH

Enhancing the physical activity levels of community-dwelling older people with frailty through an exercise intervention with or without a wearable activity tracker (WAT)-based intervention: a feasibility and pilot study

Principal Investigator: Dr. Justina Yat Wa LIU, Co-Principal Investigator: Dr. Xue BAI Co-Investigator: Dr. Paul LEE, Rick KWAN, Judy SIU

| I<br>Justina Yat Wa LIU. | hereby consent to participate | n the captioned research conduc | ted by Dr. |
|---|---|---|---|
| | cy will be retained, i.e. my perso | ay be used in future research and onal details will not be revealed a | - |
| • | the attached information sheet hicipation in the project is volunt | as been fully explained. I unders<br>ary. | stand the benefits |
| • | he right to question any parts of any time without penalty of any | the interview and/or conversatio kind. | n and can |
| Participant: | | | |
| Name of Participant | Signature | Date | |
| Researcher: | | | |
| Name of Researcher | Signature | <br>Date | |





## INFURMATION SHEET

Enhancing the physical activity levels of community-dwelling older people with frailty through an exercise intervention with or without a wearable activity tracker (WAT)-based intervention: a feasibility and pilot study

Principal Investigator: Dr. Justina Yat Wa LIU, Co-Principal Investigator: Dr. Xue BAI Co-Investigator: Dr. Paul LEE, Rick KWAN, Judy SIU

You are being invited to take part in this research project. This research project aims to investigate the effects of a wearable activity tracker (WAT)-based exercise programme on enhancing the physical activity levels among community dwelling pre-frail and frail older people.

If you decide to be in this study, your socio-demographic data will be obtained for research and education purpose. Each participating centre will be randomized to either the WAT group or the control group. The WAT group will receive a 3-month WAT-based exercise training programme (12 sessions) in addition to face-to-face and telephone support for behavioural change techniques (BCTs) and technical issues (7 sessions). Then, you will be requested to use the WAT on your own for another 3 months during the follow-up period. The control group will receive a 3-month exercise training programme without a WAT in addition to face-to-face and telephone support for BCTs.

To further understand the acceptability of the WAT intervention, all participants in the WAT group will be invited to attend a focus group interview. Your responses to interview questions will be kept confidential.

The researcher will conduct face-to-face interview and physical assessments before the programme begins, at 1 week, 1 and 3 months after the programme. The assessments include socio-demographics, 30-second chair stand test (30-s CST), Timed Up and Go test (TUG), 2-minute walk test (2MWT), 9-item Chinese Self-Efficacy for Exercise scale (CSEE), Fried Frailty Index (FFI), Physical Activity Scale for Elderly-Chinese (PASE-C), Chinese Global Physical Activity Questionnaire (C-GPAQ) and Chinese Behavioural Regulation in Exercise Questionnaire (C-BREQ-2).

Adverse events such as muscle tiredness may arise during the exercise programme. Therefore, the potential adverse events relating to the intervention and information on exercising safely will be discussed with you. All information related to you will remain confidential, and will be identifiable by codes only known to the researcher. The collected data may be used for future studies, education and academic purposes.

You have every right to withdrawn from the study before or during the study without penalty of any kind.

If you would like to know more details of this study, please contact Dr Justina Liu at 2766-4097.

If you have any complaints about the conduct of this research study, please do not hesitate to contact Ms Cherrie Mok, Secretary of the Human Subjects Ethics Sub-Committee of The Hong Kong Polytechnic University in writing (c/o Research Office of the University) stating clearly the responsible person and department of this study.

Thank you for your interest in participating in this study.

Dr. Justina Yat Wa LIU Principal Investigator